CLINICAL TRIAL: NCT03263832
Title: Demonstration of Clinical Value of Antibiofilmogramme Test for Monomicrobial S. Aureus Orthopaedic Device-Related Infection
Brief Title: Evaluation of the Antibiofilmogramme Test During Orthopaedic Device-Related Infection
Acronym: BJIBiofilm
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: BioFilm Control (Industry)
Collaborators: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 2015-A0022472
Record Dates: First submitted 2017-08-23; First posted 2017-08-28 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-03

CONDITIONS: Prosthetic Joint Infection; Staphylococcus Aureus; Biofilm
Keywords: Antibiogramme; Antibiofilmogramme
MeSH Terms: conditions — Staphylococcal Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples Without DNA — The S. aureus strains isolated will be maintained in a collection for future ancillary studies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Exposed: Patients with a monomicrobial S. aureus orhtopaedic device-related infection who have received antibiotherapy able to prevent biofilm formation following surgical intervention (from day 0 to day 7).
  Upon inclusion, antibiograms were performed on the S. aureus isolated as part of routine procedure. S. aureus isolates was further analysed via an Antibiofilmogramme, which is an experimental element added by this research.
  Interventions: Diagnostic Test: Antibiofilmogramme
- Not Exposed: Patients with a monomicrobial S. aureus orhtopaedic device-related infection who not have received antibiotherapy able to prevent biofilm formation following surgical intervention (from day 0 to day 7).
  Upon inclusion, antibiograms were performed on the S. aureus isolated as part of routine procedure. S. aureus isolates was further analysed via an Antibiofilmogramme, which is an experimental element added by this research.
  Interventions: Diagnostic Test: Antibiofilmogramme

INTERVENTIONS:
Diagnostic Test: Antibiofilmogramme — An Antibiofilmogramme (BioFilm Control) evaluates the capacity of a series of antibiotics to inhibit the growth of bacterial biofilms for a given bacterial isolate.

SUMMARY:
This is an observational study that does not change routine care.

The primary objective of this study is to investigate the correlation between the administration of an antibiotherapy able to prevent biofilm formation according to the results of the Antibiofilmogramme test, and the relapse of the infection for patient with orthopaedic device-related infection.

DETAILED DESCRIPTION:
The secondary objectives are:

A. Investigate the role of antibiogram-antibiofilmogramme concordance (in terms of S. aureus strains and prescribed antibiotics) in orthopaedic device-related infection management.

B. Investigate the capacity of S. aureus isolates to form biofilm in presence/absence of antibiotics.

C. Create an S. aureus strain collection for future ancillary studies

ELIGIBILITY:
Inclusion Criteria:

* The patient must have been informed and received a non-opposition consent form
* Patient with a monomicrobial S. aureus bone and joint infections
* Patient with prosthetic or orthopaedic device

Exclusion Criteria:

* Bone and joint infection from pressure ulcer, vascular injury or diabetic foot ulcer
* Polymicrobial prosthetic joint infection
* The patient is participating in, or has participated in within the past 3 months, another interventional study, or is currently in an exclusion period determined by a preceding study
* Patient is under judicial protection, under tutorship or curatorship
* The patient expresses his opposition to participate to the study
* It is impossible to correctly inform the patient
* The patient is pregnant, parturient or breastfeeding
* Emergency situation precluding correct study implementation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is composed of patient with a monomicrobial S. aureus orthopaedic device-related infections.
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Success or treatment failure | From surgical intervention to one year after the end of antimicrobial therapy.
  Presence or absence of microbiological treatment failure confirmed by S. aureus positive clinical samples. The diagnostic of a S. aureus positive clinical sample indicated a treatment failure. Treatment success corresponded to an absence of clinical or microbiological treatment failure, or treatment failure with positive clinical sample other than S. aureus.

OTHER OUTCOMES:
Age | Baseline (Day 0)
  (years)
Sex | Baseline (Day 0)
  (m/f)
Body mass index | Baseline (Day 0)
  (kg/m²)
Charlson Comorbidity Index | Baseline (Day 0)
  (0-37)
Localization of the infection | Baseline (Day 0)
  Knee, Hip or other
Orthopaedic device | Baseline (Day 0)
  Prothesis, screw, plate or other
Time of onset of symptoms | Baseline (Day 0)
  (date)
Time of microbiological diagnostics | Baseline (Day 0)
  (date)
Time of implantation of the device | Baseline (Day 0)
  (date)
Microbiological analysis | Baseline (Day 0)
  Number of positive S. aureus biopsy samples
Antibiogram results | Baseline (Day 0)
  Qualitative results per antibiotic type and dose: classification as sensitive, intermediate, resistance and MIC estimation by the Vitek
Surgical Therapy | Baseline (Day 0)
  Conservative treatment (arthrotomy, debriedment, synovectomy) or removal of implant (one stage, two stage)
Antibiotics taken | through study completion, an average of 1 year
  Name of the molecule, dose and duration

CONTACTS AND LOCATIONS:
Overall Officials: Frederic Laurent, PharmD - PhD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hospices Civils de Lyon, Lyon, France